CLINICAL TRIAL: NCT06703359
Title: Evaluation of the Predictive Properties of the 6-Minute Stepper Test for Long-term Mortality in Patients with COPD
Brief Title: Predictive Properties of the 6-Minute Stepper Test for Mortality in COPD
Acronym: SixSTeM-COPD
Status: Recruiting | Type: Observational
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: SixSTeM-COPD
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: COPD
Keywords: COPD; Six-minute stepper test; Pulmonary rehabilitation; Exercise testing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD referred for pulmonary rehabilitation.: Included participant were referred for pulmonary. During their baseline assessment, they performed the 6-Minute Stepper Test and were then followed for 5 years.

SUMMARY:
Retrospective study aimed to answer the following research questions :

* What are the predictive properties of the 6-minute stepper in COPD for 2-year mortality in individuals with COPD ?
* What are the predictive properties of the 6-minute stepper in COPD for 5-year mortality in invididuals with COPD ?

DETAILED DESCRIPTION:
Method: retrospective study with external validation.

The medical records of all patients referred for pulmonary rehabilitation at ADIR Association, France, between 2015 and 2023 will be screened for eligibility. Demographic data and performance during the 6-Minute Stepper Test will be collected directly from the patients' medical records.

Collected data include: age, weight, height, body-mass index, sex, long-term oxygen therapy, long-term non-invasive ventilation, oxygen uptake (from cardiopulmonary exercise testing), peak power output (from cardiopulmonary exercise testing), pulmonary function testing, disease stage according to the Global Initiative for Chronic Obstructive Lung Disease classification, modified Medical Research Council dyspnea score, smoking status, quality of life, number of disease exacerbations prior to the pulmonary rehabilitation program, number of pulmonary rehabilitation programs performed during the follow-up period, and performance during the 6-Minute Stepper Test.

Vital status (alive or deceased) will be collected from the database of the French National Institute of Statistics and Economic Studies (INSEE): https://arbre.app/insee. This variable will be collected during the first quarter of 2025.

A receiver operator curve analysis will be performed to determine the statistical threshold value (number of steps) with the best sensitivity and specificity for predicting all-cause mortality at 2 and 5 years.

Patients will then be divided into two groups based on the established threshold, and a Cox regression model will be used to determine the hazard ratio for mortality at 2 and 5 years.

Invidiual participant data from a prospective study will be used to assess the external validity of established thresholds.(https://pubmed.ncbi.nlm.nih.gov/27216848/).

Statistical analysis :

Continuous data will be expressed as mean (standard deviation), median (interquartile range), and categorical data as number (percentage). The distribution of data will be assessed using the Shapiro-Wilk test.

To determine the statistical threshold value of the 6-Minute Stepper Test with the best sensitivity and specificity for 2-year and 5-year mortality, receivor operator curves (95% confience interval) will be generated.

Patients will then be divided into two groups (based on the threshold value). The characteristics of the two groups will be compared using Fisher's exact test (categorical data), the independent Student's t-test (parametric data), or the Mann-Whitney U test (non-parametric data).

A Cox proportional hazards regression model will be used to calculate the "crude" and "adjusted" hazard ratio (95% confidence interval) for 2-year and 5-year mortality. The adjusted model will include the following variables: sex, age, FEV1 (L), modified Medical Research Council dyspnea score, BMI. Sensitivity analysis will be porformed adding smoking status, long term oxygen use and number of pulmonary rehabilitation during the follow-up.

The external validity of the model will be assessed using individual pariticipant data from a previously published study (https://pubmed.ncbi.nlm.nih.gov/27216848/).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Covered by a social security scheme;
* COPD (all stages);
* Referred for pulmonary rehabilitation;
* Completed a 6-Minute Stepper Test at the start of their program.

Non-inclusion Criteria:

* Patients under guardianship or legal supervision;
* Pregnant or breastfeeding women.

Exclusion Criteria:

* Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with COPD referred for pulmonary rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Two-year mortality | From the 6-Minute Stepper Test to two years thereafter
  Vital status (alive or deceased) will be collected from the database of the French National Institute of Statistics and Economic Studies (INSEE): https://arbre.app/insee.
Five-year mortality | From the 6-Minute Stepper Test to five years thereafter
  Vital status (alive or deceased) will be collected from the database of the French National Institute of Statistics and Economic Studies (INSEE): https://arbre.app/insee.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Bonnevie, PhD, Principal Investigator — ADIR Association
Locations (1):
- ADIR Association, Rouen, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonnable request for research purpose after publication. Request should be send to t.bonnevie@adir-hautenormandie.com
Time Frame: Data will be made available after publication.
Access Criteria: Data will be made available upon request to t.bonnevie@adir-hautenormandie.com